CLINICAL TRIAL: NCT01861171
Title: Effect of Green Tea on Adiposity, Metabolic Profile, Blood Pressure and Endothelial Function in Obese Pre-hypertensive Women
Brief Title: Effect of Green Tea in Obese Pre-hypertensive Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Antonio Felipe Sanjuliani, Prof. Dr., Rio de Janeiro State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: clinex01
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Obese; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Crossover randomized controlled double-blinded trial. Twenty women with obesity and pre-hypertension, aged 28-59 years, with stable body weight were randomized to receive a daily supplement of 3 capsules that contained either 500mg of green tea extract (GTE) or a matching placebo for 4 weeks, with a washout period of 2 weeks between the treatments.
  Interventions: Dietary Supplement: Green Tea
- Green Tea (Active Comparator): Crossover randomized controlled double-blinded trial. Twenty women with obesity and pre-hypertension, aged 28-59 years, with stable body weight were randomized to receive a daily supplement of 3 capsules that contained either 500mg of green tea extract (GTE) or a matching placebo for 4 weeks, with a washout period of 2 weeks between the treatments.
  Interventions: Dietary Supplement: Green Tea

INTERVENTIONS:
Dietary Supplement: Green Tea — Twenty women with obesity and pre-hypertension, aged 28-59 years, with stable body weight were randomized to receive a daily supplement of 3 capsules that contained either 500mg of green tea extract (GTE) or a matching placebo for 4 weeks, with a washout period of 2 weeks between the treatments.

SUMMARY:
The purpose of this study is to evaluate the effects of green tea on body weight, waist circumference, metabolic profile, inflammation, blood pressure and endothelial function in obese pre-hypertensive women.

DETAILED DESCRIPTION:
Crossover randomized controlled double-blinded trial. Twenty women with obesity and pre-hypertension, aged 28-59 years, with stable body weight were randomized to receive a daily supplement of 3 capsules that contained either 500mg of green tea extract (GTE) or a matching placebo for 4 weeks, with a washout period of 2 weeks between the treatments. Endothelial function was evaluated by peripheral arterial tonometry method, using Endo-PAT 2000®.

ELIGIBILITY:
Inclusion Criteria:

pre-hypertensive women obese adult

Exclusion Criteria:

pregnant smoker elderly

Ages: 28 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduction of blood pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lívia P Nogueira, Principal Investigator — Pedro Ernesto Universitary Hospital
Locations (1):
- Pedro Ernesto Hospital Universitary, Rio de Janeiro, Rio de Janeiro, Brazil